CLINICAL TRIAL: NCT05464719
Title: A Phase II Study of Loncastuximab Tesirine as Consolidation Strategy in Patients With LBCL in PR After CAR T-cell Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0147; NCI-2022-05750 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-07-11; First posted 2022-07-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Large B-cell Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Loncastuximab Tesirine (Experimental): Participants will receive Loncastuximab Tesirine (lonca) by vein.
  Interventions: Drug: Loncastuximab Tesirine

INTERVENTIONS:
Drug: Loncastuximab Tesirine — Given by IV
  Other Names: Lonca

SUMMARY:
To learn if loncastuximab tesirine (called "lonca" in this informed consent form) can help to control large B-cell lymphoma that is relapsed or refractory after receiving CAR T-cell therapy. The safety and possible effects of the study therapy will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

-To evaluate the efficacy of lonca as consolidation therapy in patients with relapsed or refractory LBCL who achieve PR after CAR T-cell therapy.

Secondary Objectives:

-To evaluate safety and tolerability of lonca as consolidation therapy in patients with relapsed or refractory LBCL who achieve PR after CAR T-cell therapy.

Exploratory Objective:

-To determine the pharmacodynamic effects and investigate biomarkers of response and resistance of this novel consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will be considered for inclusion in this study if they meet the following criteria:

1. Relapsed or refractory diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma, transformed indolent B-cell lymphomas and high-grade B-cell lymphoma
2. Receive standard of care treatment with an FDA-approved anti-CD19 autologous CAR T-cell product, outside of a clinical trial
3. ≥ 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
5. Achievement of PR according to Lugano 2014 response criteria 30 days after CAR T-cell therapy
6. At least 30 days must have elapsed since CAR T-cell therapy infusion
7. No evidence of CD19 expression after CAR T-cell therapy infusion is required for enrolment
8. No additional anti-tumoral therapy, with the exclusion of palliative radiotherapy, must have been received after CAR T-cell therapy
9. Absolute neutrophil count (ANC) of ≥ 1.0×109/L without growth factor support for 3 days prior to screening assessment.
10. Platelet count of ≥ 50×109/L without transfusion for 3 days prior to screening assessment.
11. Creatinine clearance (as estimated by Cockcroft Gault) ≥ 30 mL/min
12. Serum alanine transaminase (ALT) or aspartate transaminase (AST) ≤ 2.5 upper limit of normal (ULN)
13. Total bilirubin ≤2 mg/dL, except in subjects with Gilbert's syndrome.
14. Cardiac ejection fraction ≥ 45% with no evidence of clinically significant pericardial effusion
15. Baseline oxygen saturation > 92% on room air
16. No evidence or suspicion of lymphoma actively involving the central nervous system (CNS)
17. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
18. Resolution of any previous CRS and/or ICANS to grade 0.

4.3 Exclusion criteria

Subjects will be ineligible for this study if they meet the following criteria:

1. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
2. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. prostate, cervix, bladder, breast) unless disease free for at least 12 months
3. History of Richter's transformation of chronic lymphocytic leukemia (CLL)
4. Treatment with CAR T-cell therapy on clinical trial as immediate treatment before enrollment
5. Prior treatment with lonca
6. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the Principal investigator
7. Known history of infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive). A history of HIV, hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
8. Subjects with active cardiac atrial or cardiac ventricular lymphoma involvement
9. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrolment
10. Primary immunodeficiency
11. History of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring active systemic immunosuppression/systemic disease modifying agents within the last 2 years
12. History of clinically significant deep vein thrombosis or pulmonary embolism within 1 month of enrollment per investigators discretion.
13. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
14. History of severe immediate hypersensitivity reaction to any of the agents used in this study
15. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the PBD on the fetus or infant.
16. Subjects of both genders who are not willing to practice birth control. Women of childbearing potential must use a highly effective method of contraception (hormonal birth control such as birth control pills, intravaginal ring, skin patch, implant or injection, intrauterine device or surgical sterilization) until 9 months after last dose of lonca, and men with female partners who are of childbearing potential should use a condom when sexually active until 6 months after the last dose of lonca
17. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation Trial Treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion to complete response | through study completion and or average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Strati, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org